CLINICAL TRIAL: NCT04670471
Title: Single-centre, Randomised, Prospective, Open-label, Three-period, Phase 1 Clinical Trial for Assessment of the Pharmacodynamic and Pharmacokinetic Interaction of Remimazolam and Remifentanil
Brief Title: Assessment of the Pharmacodynamic and Pharmacokinetic Interaction of Remimazolam and Remifentanil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Paion UK Ltd. (Industry)
Collaborators: University Medical Center Groningen (Other); QPS Holdings LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: CNS7056-025; 2020-003806-30 (EudraCT Number)
Record Dates: First submitted 2020-11-25; First posted 2020-12-17 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Anesthesia
MeSH Terms: interventions — remimazolam; Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Remimazolam + Remifentanil plasma concentration of 2.0 ng/mL (Experimental): Each participant will receive study medication on three different occasions:
  Session 1: remimazolam alone Session 2: remimazolam plus remifentanil 0.5 ng/mL Session 3 : remimazolam plus reminfentanil 2.0 ng/mL During each session remimazolam will be dosed in a step-up / step-down manner while the remifentanil target concentration will be kept constant.
  Interventions: Drug: Remimazolam; Drug: Remifentanil
- Remimazolam + Remifentanil plasma concentration of 4.0 ng/mL (Experimental): Each participant will receive study medication on three different occasions:
  Session 1: remimazolam alone Session 2: remimazolam plus remifentanil 0.5 ng/mL Session 3 : remimazolam plus reminfentanil 4.0 ng/mL During each session remimazolam will be dosed in a step-up / step-down manner while the remifentanil target concentration will be kept constant.
  Interventions: Drug: Remimazolam; Drug: Remifentanil
- Remimazolam + Remifentanil plasma concentration of 0.1 ng/mL (Experimental): Each participant will receive study medication on three different occasions:
  Session 1: remimazolam alone Session 2: remimazolam plus remifentanil 0.5 ng/mL Session 3 : remimazolam plus reminfentanil 0.1 ng/mL During each session remimazolam will be dosed in a step-up / step-down manner while the remifentanil target concentration will be kept constant.
  Interventions: Drug: Remimazolam; Drug: Remifentanil
- Remimazolam + Remifentanil plasma concentration of 1.0 ng/ml (Experimental): Each participant will receive study medication on three different occasions:
  Session 1: remimazolam alone Session 2: remimazolam plus remifentanil 0.5 ng/mL Session 3 : remimazolam plus reminfentanil 1.0 ng/mL During each session remimazolam will be dosed in a step-up / step-down manner while the remifentanil target concentration will be kept constant.
  Interventions: Drug: Remimazolam; Drug: Remifentanil

INTERVENTIONS:
Drug: Remimazolam — Remimazolam is an intravenous anaesthetic and sedative drug. Remimazolam exhibits its anaesthetic effects via the benzodiazepine binding site at the GABAA receptor.
  Other Names: Byfavo, CNS7056
Drug: Remifentanil — Remifentanil is a commonly used opioid in anaesthetic practice. It is a potent and fast-acting analgesic.
  Other Names: Ultiva

SUMMARY:
This trial is designed to quantify the pharmacodynamic (PD) and pharmacokinetic (PK) interaction(s) between an anaesthetic drug (remimazolam) and an opioid (remifentanil). Remimazolam is a new anaesthetic drug with a sedative effect, which, in combination with an opioid can be used to achieve general anaesthesia. To date, however, no clinical trials have been conducted to specifically assess the potential for drug-drug interactions between remimazolam and remifentanil. Greater understanding of the potential for such interactions will help define more appropriate dosing regimens with less over-sedation and associated side effects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adults ≥18 to ≤70 years old
* American Society of Anesthesiologists (ASA) Physical Status 1
* Body mass index (BMI) >18 to <30 kg/m2
* Bilateral patent a. radialis
* For female volunteers of childbearing potential: Negative results of 2 pregnancy tests, the first test taken at the start of Screening and the second test taken from the morning urine within 3 hours before the start of the administration of the IMP as well as consent to use highly effective birth control from the last menstrual cycle prior to the start of the IMP until the end of the trial follow-up procedures. Highly effective methods of birth control include:

  * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral/intravaginal/transdermal)
  * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral/injectable/implantable)
  * Intrauterine device (IUD)
  * Intrauterine hormone-releasing system (IUS)
  * Bilateral tubal occlusion
  * Vasectomised partner (provided that the partner is the sole sexual partner of the female patient of childbearing potential and that the vasectomised partner has received medical assessment of the surgical success).
  * Sexual abstinence

Women who had their last menstruation at least two years ago or who underwent surgical interventions (surgical birth control, bilateral oophorectomy, hysterectomy, etc.) are regarded as having no childbearing potential.

* For male participants, their partner must not become pregnant during the trial. They should inform their partner about this. They must also agree to use of barrier methods of contraception during the trial.
* Subject agrees not to use alcohol for 2 days, not to use nicotine for 1 week, and not to use recreational drugs for 2 weeks prior to the first period until End of Trial
* Understanding of the trial procedures and be willing to follow the instructions of the Investigator or centre staff during the course of the clinical trial
* Written informed consent obtained from the subject

Exclusion Criteria:

* Known intolerance to benzodiazepines, flumazenil, opioids or any ingredients of the remimazolam drug products (e.g., dextran, lactose)
* Pregnancy, or currently breastfeeding
* Have current neurological disorder(s) (epilepsy, the presence of a brain tumour, a history of brain surgery, hydrocephalic disorders, depression needing treatment with anti-depressive drugs, a history of brain trauma, a subarachnoidal bleeding, TIA or cerebral infarct, psychosis or dementia, schizophrenia, alcohol or drug abuse).
* Have a disease(s) involving the cardiovascular system (hypertension, coronary artery disease, prior acute myocardial infarction, any valvular and/or myocardial disease involving decrease in ejection fraction, arrhythmias, which are either symptomatic or require continuous medication/pacemaker/automatic internal cardioverter defibrillator)
* Recent (<3 months) use of psycho-active medication (benzodiazepines, anti-epileptic drugs, Parkinson's medication, neuroleptics, anxiolytics, anti-depressant drugs, and opioid analgesics)
* A history of illicit drug or alcohol abuse within two years prior to screening
* Any ongoing condition considered by the Investigator as potentially relevant to the trial
* Any medical history considered by the Investigator as potentially relevant to the trial
* An employee or direct relative of an employee of the trial site, the CRO or the Sponsor.
* Resting HR <45 bpm or ≥90 bpm OR resting SABP <90 mmHg or ≥140 mmHg OR resting DABP <50 mmHg or ≥90 mmHg, except for those cases where hypertension is accompanied by tachycardia as judged by the screening physician.
* Positive urine drug screening test (amphetamines, methamphetamines, benzodiazepines, barbiturates, marijuana, cocaine, and opioids).
* Positive Covid-19 screening test
* Any participant as judged by the PI or Sub-Investigator to be inappropriate for the trial for any other reason
* Clinically significant, as judged by the Investigator abnormal ECG
* Clinically significant abnormal laboratory values
* Participation in a clinical trial of an Investigational Drug or Medical Device within three months prior to the Screening Visit
* Blood donation of ≥500mL within three months prior to Screening Visit
* Prior participation in this clinical trial. However, non-dosed drop-outs can participate in the trial again but will need to be re-screened.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Exposure-response model describing the relationship between effect-site concentrations of remimazolam and plasma concentrations of remifentanil and MOAA/S corresponding to mild, moderate and deep sedation. | Through study completion, approximately 3 weeks

SECONDARY OUTCOMES:
Exposure-response model describing the relationship between effect-site concentrations of remimazolam and plasma concentrations of remifentanil and BIS corresponding to mild, moderate and deep sedation. | Through study completion, approximately 3 weeks
Performance characteristics for the TCI models used (remimazolam and remifentanil) according to Varvel et al. These include median absolute performance error, median performance error, wobble and divergence. | Through study completion, approximately 3 weeks
Exposure response models for tolerance to laryngoscopy | Through study completion, approximately 3 weeks
Exposure response models for tolerance to tetanic stimulus | Through study completion, approximately 3 weeks
Exposure response models for BIS | Through study completion, approximately 3 weeks
Exposure response models for hemodynamic alterations in terms of heart rate, arterial blood pressure (ABP), mean arterial pressure (MAP), stroke volume and cardiac output | Through study completion, approximately 3 weeks
Exposure response models for respiratory depression | Through study completion, approximately 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Remco Vellinga, MD, Principal Investigator — University Medical Center Groningen (UMCG)
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Varvel JR, Donoho DL, Shafer SL. Measuring the predictive performance of computer-controlled infusion pumps. J Pharmacokinet Biopharm. 1992 Feb;20(1):63-94. doi: 10.1007/BF01143186. PMID 1588504
- [Derived] Vellinga R, Koomen JV, Eleveld DJ, Stohr T, Pesic M, Struys MMRF, Colin PJ. Influence of Remifentanil on the Pharmacokinetics and Pharmacodynamics of Remimazolam in Healthy Volunteers. Anesthesiology. 2025 Apr 1;142(4):666-679. doi: 10.1097/ALN.0000000000005348. Epub 2025 Jan 15. PMID 40067039